CLINICAL TRIAL: NCT00882375
Title: Efficacy and Safety Following Use of a Novel Nicotine Replacement Therapy. A Multicenter, Randomized, Double Blind, Placebo Controlled, Parallel Group, 52 Week Study in Smokers Motivated to Quit.
Brief Title: Efficacy and Safety Following Use of a Novel Nicotine Replacement Therapy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: McNeil AB (Industry)
Responsible Party: Sponsor
Organization: Johnson & Johnson Consumer and Personal Products Worldwide (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6431111; 2008-006845-13 (EudraCT Number)
Record Dates: First submitted 2009-04-15; First posted 2009-04-16 (Estimated); Last update posted 2012-07-02 (Estimated); Status verified 2012-06

CONDITIONS: Smoking Cessation
Keywords: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation | interventions — Nicotine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Nicotine (Experimental): Nicotine
  Interventions: Drug: Nicotine
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Nicotine — Nicotine administered using novel NRT user instructions
  Other Names: NRT
  Arms: Nicotine
Drug: Placebo — Placebo administered using novel NRT user instructions
  Arms: Placebo

SUMMARY:
A comparison of a novel nicotine replacement therapy and placebo treatment in smokers motivated to quit smoking.

DETAILED DESCRIPTION:
Efficacy and safety study following use of a novel nicotine replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older male and female cigarette smokers motivated and willing to stop smoking
* Female participants of child-bearing potential should use a medically acceptable means of birth control.
* Evidence of a personally signed and dated informed consent document indicating that the subject has been informed of all pertinent aspects of the study and consents to participate.

Exclusion Criteria:

* Unstable angina pectoris or myocardial infarction during the previous 3 months.
* Pregnancy, lactation or intended pregnancy (non-pregnancy will be verified by urine pregnancy test for female participants of child-bearing potential).
* Participation in other clinical trials within the previous three months and during study participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 479 (Actual)
Dates: Start 2009-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Self-reported continuous abstinence from smoking verified by exhaled CO levels of less than 10 ppm. | at weeks 2, 6, 24 and 52

SECONDARY OUTCOMES:
Self-reported continuous abstinence from smoking, verified by exhaled CO levels of less than 10 ppm. | weeks 2, 4, 8, 12, 16, and 20
Self-reported 7-day point prevalence abstinence from smoking verified by exhaled CO levels of less than 10 ppm. | weeks 4, 6, 8, 12, 16, 20, 24, and 52
Ratings of craving/urge to smoke and withdrawal symptoms. | baseline to 24 weeks
Cotinine levels in saliva. | baseline, and weeks 2, 6, 12 and 24
Product acceptability | weeks 1, 6 and 12

CONTACTS AND LOCATIONS:
Overall Officials: Elisabeth Kruse, PhD, Study Director — McNeil AB
Locations (3):
- Gentofte University Hospital, Hellerup, Denmark
- Germany (2):
  - University of Heidelberg, Mannheim
  - University Hospital of Tuebingen, Tübingen

REFERENCES:
- [Derived] Roche F, Pepin JL, Achour-Crawford E, Tamisier R, Pichot V, Celle S, Maudoux D, Chouchou F, Ntougou-Assoumou HG, Levy P, Barthelemy JC; PROOF Study Group. At 68 years, unrecognised sleep apnoea is associated with elevated ambulatory blood pressure. Eur Respir J. 2012 Sep;40(3):649-56. doi: 10.1183/09031936.00162710. Epub 2012 Apr 20. PMID 22523363